CLINICAL TRIAL: NCT05175729
Title: Comparing Anterior Segment Parameters During Pregnancy and Post-Pregnancy
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Çisil Erkan Pota, Medical Doctor, Akdeniz University
Other Study IDs: Study 2
Record Dates: First submitted 2021-12-01; First posted 2022-01-04 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Pregnancy Related
Keywords: Pregnancy; Anterior segment; Corneal Topography; Biometry
MeSH Terms: interventions — Corneal Topography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant Group: First trimester pregnant group would be included and will be followed up in second, third trimesters and after pregnancy
  Interventions: Diagnostic Test: Comprehensive Ophthalmologic Examination
- Control group: Age-, sex-matched healthy volunteers
  Interventions: Diagnostic Test: Comprehensive Ophthalmologic Examination

INTERVENTIONS:
Diagnostic Test: Comprehensive Ophthalmologic Examination — Measurements of best-corrected visual acuity, refractive error, intraocular pressure, axial length, slit lamp examination of the anterior segment, dilated fundus examination, and anterior segment parameters,corneal topography
  Other Names: Corneal Topography; Biometry; Auto refractometry; Non contact tonometry

SUMMARY:
The aim of this study is to evaluate anterior segment changes during and after pregnancy, and compare them with non pregnant healty women

DETAILED DESCRIPTION:
Pregnancy is a physiological process in which many systems such as cardiovascular, pulmonary, renal, hematological and visual systems are affected, especially the endocrine system. Many organs, including the eye and orbit, are affected by the physiological interaction between the fetus and the mother. In most pregnant women, these effects are at the physiological level and are temporary; Sometimes it can be pathological and permanent. Hormonal, coagulative and hemodynamic changes are responsible for most of the ocular adaptations. Changes in corneal curvature, sensitivity and thickness are observed during pregnancy. It has been reported that corneal curvature increases with pregnancy, this increase occurs in the last trimester and returns to first trimester values at the end of the breastfeeding period. Although the etiology of this steepening of the cornea has not been clearly clarified, it is thought that it may be due to corneal edema caused by hormonal changes. However, it's not recommended for pregnant women to prescribe contact lenses because their variable keratometric values. A decrease in corneal sensitivity during pregnancy has been detected by esthesiometry in many studies. It decreases especially in the third trimester and returns to normal around the 2nd month after delivery. The corneal thickness measured by pachymeter may increase in pregnant women. some of them had myopic shift. In a study, 83 pregnant women were examined to determine the causes of visual disturbances during pregnancy and postpartum period. Previous studies reported that there was a change in favor of myopia (-0.9±0.3D) during pregnancy and it returned to pre-pregnancy levels in the postpartum period. Unstable refractions were thought to be due to changes in corneal thickness and curvature.

As a result, it was stated that the refractive change was temporary and in favor of myopia. It is recommended to wait up to several weeks postpartum before prescribing new eyeglasses [8].

There are various reports about IOP in normal pregnant women. In most of these studies, a decrease was found in IOP during pregnancy. In a prospective study, a decrease in IOP was found in the second and third trimesters of pregnancy, and it was shown that this change returned in the first month postpartum.

Before planning an anterior segment surgeries such as cataract and refractive surgery, changes in pregnancy should be taken into account and attention should be paid to surgical timing. The aim of this study is to reveal whether there is a change in anterior segment parameters in pregnancy period

ELIGIBILITY:
Inclusion Criteria:

* Ages between 20-40 years
* Pregnant women with a gestational age less than 14 weeks in the first examination
* Having no systemic disease before and during pregnancy
* Having a spherical refractive error of less than 4 diopters, and/or had a cylindrical refractive error of less than 2 diopters

Exclusion Criteria:

* Having systemic disease, having ocular pathology that may decrease visual acuity
* Usage of systemic drugs or topical ocular drops
* Usage of exogenous hormones and entered menopause

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnancy
Study Population: Pregnan women in their first pregnancy will be followed-up during pregnancy period (first, second, third trimesters) and post partum period.
  Healthy age-, sex- matched control group will be used to compare
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Corneal thickness | 40 weeks
  Corneal thickness in mikrometer value
Anterior chamber volume | 40 weeks
  Anterior chamber volume in mm3
Anterior chamber depth | 40 weeks
  Anterior chamber depth in mm
Anterior chamber angle | 40 weeks
  Anterior chamber angle in degree
Lens power | 40 weeks
  in diopters
Anterior flat keratometry | 40 weeks
  in Diopters
Steep keratometry | 40 weeks
  in Diopters
Mean keratometry | 40 weeks
  in Diopters
Tonometry | 40 weeks
  İntraocular pressure measurement in mmHg
Best corrected visual acuity assessment | 40 weeks
  Snellen and logMAR chart
Blood pressure measurement | 40 weeks
  Systemic blood pressure
Auto refractometer | 40 weeks
  Refractive error measurement in diopter
Axial length | 40 weeks
  Axial length in mm

CONTACTS AND LOCATIONS:
Overall Officials: Çisil Erkan Pota, MD, Principal Investigator — Akdeniz University Hospital
Locations (1):
- Akdeniz University Hospital, Antalya, Konyaaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No